CLINICAL TRIAL: NCT04199429
Title: Relationship-based Care Model in Pediatrics: a Randomized Controlled Trial to Implement the Parents' Perception of Quality of Nursing Care
Brief Title: Relationship-based Care Model in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Urbino "Carlo Bo" (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Davide Sisti, Principal Investigator, University of Urbino "Carlo Bo"
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UniUrb
Record Dates: First submitted 2019-12-02; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Depression, Anxiety; Nurse-Patient Relations
Keywords: Relationship-based care; Pediatric; Caregiver anxiety; Nurse job satisfaction; Nurse
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Each nurse applied the RBC model through the treatment "Take 5 minutes" (T5M), to parents allocated to the experimental group. This consisted in devoting some time (from 5 to 10 minutes) to improving the relationship with the parent. This treatment can be considered as the practical development of the core principles of the RBC model by the study team.
  During the T5M the nurse applied the strategies of empathic communication and active listening, learned during the education and training phase. The treatment lasted from 5 to 10 minutes and was delivered once per day during the admission of the patient.
  The T5M time was considered as additional or supplementary, but not substitutive, of the standard nursing time dedicated daily to patients and parents.
  Interventions: Behavioral: Relationship-Based Care
- Control (Active Comparator): Standard nursing time dedicated daily to patients and parents.
  Interventions: Behavioral: Relationship-Based Care

INTERVENTIONS:
Behavioral: Relationship-Based Care

SUMMARY:
Aim: To evaluate whether the application of the Relationship-based Care (RBC) model as a treatment called "Take 5 minutes" (T5M) affects the level of anxiety and depression of the parent, the level of the parent perceived quality of nursing care and the work satisfaction of the nursing staff.

Design: Single-blind randomized controlled trial.

Methods: The trial was performed from February to July 2016. The trial was conducted with one intervention (N=101) and one control group (N=90). Nurses applied the RBC model as a treatment, named "Take 5 Minutes", that consisted of dedicating some short time (from 5 to 10 minutes) to the relationship with the parents, using specifically designed communication strategies. The primary outcome was the evaluation of anxiety and depression of parents, the secondary was the parent perceived quality of nursing care.

ELIGIBILITY:
Inclusion Criteria:

* the parents of the children admitted to two Pediatric Units in a nationally renowned university hospital in the North-East of Italy
* had knowledge of the Italian language spoken and written
* were available for participation in the study by signing the informed consent

Exclusion Criteria:

* Parents of hospitalized patients for a duration of less than 4 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from T0 to T1 and T2 of the Hospital Anxiety and Depression Scale (HADS) scores | T0: admission of the patient; T1: 4th day after the admission; T2: at discharge (expected mean value = 6.2 days after admission [standard deviation = 2.0])
  The Hospital Anxiety and Depression Scale (HADS) has been used to determine the anxiety and depression of the parents of hospitalized children. HADS is a fourteen items scale (seven items related to anxiety and seven to depression): each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. A cut-off point of 8/21 for anxiety or depression has been previously established in the literature.

SECONDARY OUTCOMES:
Caring Behaviors Inventory (CBI) | T2: at discharge of the patient (expected mean value = 6.2 days after admission [standard deviation = 2.0])
  The Caring Behaviors Inventory (CBI) was used to assess the quality of nursing care perceived by the parents. CBI has 24-items, divided into four dimensions: presence, compliance, competence, and care; each item is a Likert-scale ranging from 0 to 4.
Change of the job satisfaction of the nurses | 6 months
  A "Job Satisfaction" questionnaire was used to measure the job satisfaction of the nurses. This questionnaire is composed by 44-items. It was assessed at the beginning (February 2016) and at the end (July 2016) of the data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Sisti, Ph.D., Principal Investigator — University of Urbino "Carlo Bo"

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Barbieri I, Sisti D, Di Falco A, Galeazzo M, Amatori S, Rocchi MBL, Perilongo G. Relationship-based care model in paediatrics: A randomized controlled trial to implement the parents' perception of the quality of nursing care. J Adv Nurs. 2020 Dec;76(12):3597-3608. doi: 10.1111/jan.14585. Epub 2020 Oct 3. PMID 33009852